CLINICAL TRIAL: NCT05960175
Title: Impact of Patient Involvement in Alerts Management of Telemonitoring CPAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asten Sante (Industry)
Collaborators: Slb Pharma (Other); Nouvéal (Unknown); Withings (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPIAM
Record Dates: First submitted 2023-07-11; First posted 2023-07-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: OSA
Keywords: OSA; Cheyne-Stokes respiration (CSR); Continuous positive airway pressure (CPAP); Telemedicine
MeSH Terms: conditions — Cheyne-Stokes Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard CPAP telemonitoring (No Intervention): Patients are treated with CPAP and the home healthcare provider carries out monitoring in line with current practice (telemonitoring of treatment and regular home visits).
- New CPAP telemonitoring approach (Experimental): Patients are treated with CPAP and the home healthcare provider is offering a new approach to remote monitoring in which patients are involved in managing their CPAP treatment using two connected devices (the Scanwatch connected watch + the mobile application Asten&masanté) in the first 4 months of treatment.
  Interventions: Device: New telemonitoring approach using 2 connected devices : Scanwatch connected watch + Asten&masanté application

INTERVENTIONS:
Device: New telemonitoring approach using 2 connected devices : Scanwatch connected watch + Asten&masanté application — The home healthcare provider will monitor the treatment remotely and make home visits, as in the control group. However, in the case of technical alerts concerning CPAP treatment (problems with observance, leaks, residual apneas), the provider will send the patient a notification via the mobile application in order to provide advice/instructions so that the patient can resolve the alert independently. The provider will monitor the resolution of alerts remotely and may contact the patient by telephone or come to your home if necessary.
  If the connected watch detects an abnormal heart rhythm at night, the patient receives a notification and can undergo an electrocardiogram.
  Arms: New CPAP telemonitoring approach

SUMMARY:
Adherence to CPAP determines the expected benefits of the treatment. A dose-benefit relationship has been demonstrated for both functional and cardiovascular benefits. The first few days' use of the device are decisive in determining long-term compliance. In this context, daily monitoring of the data teletransmitted means that we can be more responsive to problems of compliance during the first few days of use; the contribution of telemonitoring can be very positive in a context of poor compliance.

In France, compulsory health insurance coverage of CPAP treatment is authorised for patients aged over 16 with clinical symptoms and an AHI ≥15 events per hour and <30 events/h in patients with severe cardiovascular co-morbidity. These patients are often not very sleepy due to sympathetic hypertonia with a shorter sleep duration. They are at high risk of non-compliance.

The IPIAM study specifically targets a population at cardiovascular risk and at high risk of non-compliance with CPAP treatment. The IPIAM study aims to involve patients in the success of their treatment via remote monitoring and to show that this approach makes it possible to improve the handling of alerts and to participate in the therapeutic support of the patient. Finally, this population also shares the risk of heart rhythm disorders. As part of a cross-disciplinary inter-pathology telemonitoring approach, it also makes sense to screen for cardiac rhythm disorders by wearing a connected watch.

DETAILED DESCRIPTION:
IPIAM is a prospective randomized controled study with two arms. Two approaches to telemonitoring will be compared: the standard telemonitoring carried out by the home healthcare provider (standard of care) will be compared with a new approach in which the patient is involved in managing his treatment by collecting vitals and notifying alerts via two connected devices (a connected watch and a mobile application).

The study will comprise 2 phases :

1. an initial interventional, comparative, randomised phase corresponding to the first 4 months of CPAP treatment,
2. an observational period with standard telemonitoring, lasting until the 12th month of treatment.

In this study, all patients will be treated with the same continuous positive airway pressure ventilator (AirSense 11 Autoset, ResMed).

CPAP alerts will be checked by the home healthcare provider's technicians every week and then managed differently depending on the randomisation group.

Each patient will be seen twice in pulmonology consultations, once for the inclusion visit and once 4 months after CPAP initation.

ELIGIBILITY:
Inclusion Criteria:

* Adult with newly diagnosed OSA (with central apnea index <5 ev/h), justifying CPAP and with low sleepiness (Epworth score <11 at inclusion).
* Patient with at least 1 cardiovascular risk factor (obesity, type I or II diabetes with or without treatment, permanent hypertension with or without treatment, heart failure with preserved ejection fraction, valve disease, history of atrial fibrillation, history of ischaemic heart disease, history of stroke).
* Patient with a smartphone and who agrees to use connected objects during the study.
* Signed informed consent form,
* Subject affiliated to a health insurance system, or is a beneficiary.

Exclusion Criteria:

* Patients already fitted with a CPAP machine,
* Patients with permanent atrial fibrillation,
* Patients whose state of health is not stable or requires heavy treatment,
* Patients with cognitive problems.
* Patients participating in another intervention research in pulmonology.
* Vulnerable subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
CPAP treatment adherence | Month 4
  Measurement of the average daily duration of use of the CPAP (expressed in hours) over the last 30 nights, 4 months after initiation of treatment. The duration of use will be compared between both groups.

SECONDARY OUTCOMES:
Quality of CPAP treatment assessed by leaks | Month 1, Month 2, Month 3, Month 4
  Measurement of the average leaks (expressed in liter per minute) per month using the daily data teletransmitted by CPAP ventilator throughout the follow-up period.
Quality of CPAP treatment assessed by apnea hypopnea index | Month 1, Month 2, Month 3, Month 4
  Measurement of the average residual apnea hypopnea index (expressed in number of event per hour) per month using the daily data teletransmitted by CPAP ventilator throughout the follow-up period.
long term CPAP treatment adherence | Month 6, Year 1
  Measurement of the average daily duration of use of the CPAP (expressed in hours) over the last 30 nights, 6 months and 1 year after initiation of treatment.
Number of nights with Cheynes Stoke Respirations (CSR) | over the first 4 months
  Average number of nights with CSR per patient per 30-day period during the first 4 months of treatment.
Nocturnal heart rate | over the first 4 months
  Night-time heart rate teletransmitted daily by the connected watch during the first 4 months, only in the experimental group.
Number of alerts | over the first 4 months
  Average number of technical and medical alerts (related to adherence, leaks, apnea, CSR, increase in heart rate, atrial fibrillation) per patient per 30-day period during the first 4 months of treatment.
Number of medical events (pneumology and cardiology consultations, hospitalizations) related to OSA | Month 4
  Average number of medical events (pneumology and cardiology consultations, hospitalizations) related to OSA per patient
F-SUS questionnaire | Month 4
  The French System Usability Scale (SUS) is a questionnaire evaluating the patient satisfaction on usability of interactive systems. The questionnaire comprises 10 questions and the score of user satisfaction varies from 0 to 100 (0 lowest score; 100 highest score).
Number of home healthcare provider interventions | over the first 4 months
  Average number of home healthcare provider interventions (phone call, home visit, remote assistance) per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Prigent, Dr, Principal Investigator — Polyclinique Saint-Laurent
Locations (11):
- France (11):
  - CH Départemental Vendée, La Roche-sur-Yon, France
  - AP-HP Hôpital Européen Georges, Paris, France
  - CHU Angers - Service de pneumologie, Angers
  - CHU Dijon-Bourgogne, Dijon
  - CH Versailles, Le Chesnay
  - CH Le Mans, Le Mans
  - CHU Nancy, Nancy
  - AP-HP Pitié Salpêtrière, Paris
  - AP-HP Bichat Claude Bernard, Paris
  - Polyclinique Saint-Laurent - Groupe médical de pneumologie, Rennes
  - CHU Rouen - Charles Nicolle, Rouen

IPD SHARING:
Plan to Share IPD: No